CLINICAL TRIAL: NCT03079128
Title: Evaluation of a Commercial Program on Weight Loss and Health Outcomes 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Renee J. Rogers, Principal Investigator, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO17010232
Record Dates: First submitted 2017-02-27; First posted 2017-03-14 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Weight Watchers Intervention
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — Weight Watchers Intervention

SUMMARY:
There is a body of evidence that has evaluated the effect of Weight Watchers, a commercially available weight loss program, on changes in body weight. The current investigation aims to add to this body of evidence by providing additional data on changes in body weight and enhance the current evidence-base in regards to evaluating other health-related outcomes.

There is little evidence that demonstrates whether or not the weight loss as a result of the Weight Watchers program elicits changes in health-related functional outcomes such as aerobic capacity, flexibility, sleep, and other psychological measures. Additionally, within a scientific research protocol, measures of adherence and satisfaction will also be evaluated evaluated. This study will evaluate these outcomes beyond weight changes achieved across the 24-week program.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ages 18-75 years. Set "soft quotas" on the number of male and female participants. The desire is to have an 80% female/20% male split.
* Willing to enroll in the Weight Watchers Program
* With or without previous Weight Watchers experience Set maximum quota on the number of participants with previous Weight Watchers experience at 65%.
* Self-reported height/weight resulting in a Body Mass Index (BMI) of 25 to 43 (will re-screen at facility).
* Self report that he/she feels the need to lose weight.
* Willing to discontinue any current over-the-counter (OTC) supplements not recommended/prescribed by physician, with the exception of multivitamins or other vitamin supplement.
* Willing to follow recommendations required by study protocol.
* Willing to include demographic information (e.g., ethnicity, income and education).
* Use of a personal iPhone on a daily basis

  1. iPhone must have iOS 8.0 or later
  2. Must have at least 600 MB of available storage to accommodate the size of the app
* The willingness and ability to navigate and use applications on their iPhone on a daily basis (minimum training will be provided)
* Reliable home Wi-Fi access
* Ability to commit to attending up to 27 study visits in approximately 26 weeks:

  1. Ability to commit (to best of their ability) to attending weekly meetings, 30-60 minutes in duration, on the same day and at the same time each week for 24 consecutive weeks.
  2. Ability to commit to up to 3 additional study visits at Weeks 0, 12 and 24, with each visit being 60-90 minutes in duration to complete assessments (height, weight, questionnaires, physical measures).

Exclusion Criteria:

* Currently, or within the last 6 months, trying to lose weight by following guidelines (e.g., self-initiated programs such as 5-2, or Atkins) or a structured weight-loss program (e.g., at a medical center, university, commercial programs)
* A member of Weight Watchers within the past 12 months.
* Involved in any other related research studies and self-report agreeing to not enroll in other studies that may affect weight or health outcomes over the next 12 months.
* Pregnant or nursing, or planning on becoming pregnant over the next 9 months.
* Weight loss of ≥ 5 kg in the previous 6 months.
* History of clinically diagnosed eating disorder.
* Reported health problems that make weight loss or unsupervised exercise unsafe or unreasonable (e.g., orthopedic limitations, heart problems)
* Untreated thyroid disease or any changes (type or dose) in thyroid medication in last 6 months.
* Taking any prescription medication with known effects on appetite or weight (e.g., oral steroids, weight loss medications such as Qysmia, Contrave, etc.) with the exception of subjects on a stable dose of Selective Serotonin Reuptake Inhibitors (SSRIs) for 6 months
* Diuretic use for hypertension over 1.5mg per day
* Chronic/inflammatory gastrointestinal disorders (irritable bowel syndrome acceptable).
* History of heart problems (e.g., angina, bypass surgery, myocardial infarction, etc.) within previous 6 months.
* Resting systolic blood pressure >160 mmHg or resting diastolic blood pressure >100 mmHg
* Diagnosis of type 1 or type 2 diabetes.
* Previous surgical procedure for weight loss.
* Major surgery within the previous 6 months.
* Presence of implanted cardiac defibrillator or pacemaker.
* History of cancer within past 5 years or current treatment for cancer (completely resected basal or squamous cell carcinoma acceptable if treatment completed more than 6 months prior to enrollment).
* Hospitalization for psychiatric problems during the past 12 months.
* Consuming more than 14 alcoholic drinks per week or not more than 3 drinks per day.
* Planning to relocate in the next 9 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2017-09-18 (Actual); Study Completion 2017-09-18 (Actual)

PRIMARY OUTCOMES:
Body Weight Change | Baseline, 3 months, and 6 months
  To examine the effect of a 24-week commercially available weight loss program on weight change.

SECONDARY OUTCOMES:
Change in Aerobic Capacity | Baseline, 3 months, and 6 months
  Aerobic Capacity: Participants will complete a 6 minute walk test on a designated walking course. The 6 minute walk test is a measure of functional and aerobic capacity. Participants will asked to walk at a brisk, yet comfortable pace for a total of 6 minutes.
Change in Flexibility | Baseline, 3 months, and 6 months
  Flexibility: Lower body flexibility will be assessed through the sit and reach test. The sit and reach is a common test to measure lower back and lower body flexibility.
Change in Sleep Quality and Duration | Baseline, 3 months, and 6 months
  Sleep quality and duration. Participants will be asked to complete the Pittsburgh Sleep Quality Index (PSQI) at baseline, Months 3 and 6. The PSQI is a validated self-report measure of sleep duration and sleep quality.
Change in Happiness | Baseline, 3 months, and 6 months
  Participants will be asked to complete the Oxford Happiness Questionnaire at baseline, Months 3 and 6. The OHQ is a validated self-report measure for broad personal happiness. Respondents rate 29 sentences on a 6 point Likert scale (1, strongly disagree; 6, strong agree).
Change in Food Cravings | Baseline, 3 months, and 6 months
  The Food Craving Inventory-II (FCI-II) is a validated self-report measure for general cravings and cravings for specific types of foods and will be completed at baseline, Months 3 and 6. Respondents rate the frequency of cravings since the last time they completed the survey for each of 33 food items using a five-point Likert scale (1, never; 2, rarely; 3, sometimes; 4, often; 5, always/almost every day). The FCI-II consists of 5 scales (sweets, high fats, carbohydrates/starches, fast food fats, and fruits & vegetables) that constitute the higher order construct of food cravings (the total score).
Program Adherence | Baseline, 3 months, and 6 months
  Data on adherence (attendance at meetings and use of the points system) will also be collected. Attendance data will be recorded by Weight Watchers staff at every meeting. These data will be confirmed by a member of the research staff that will be attending the weekly Weight Watchers meetings. In addition, the weekly weights obtained at the intervention sessions will be provided to the investigators by the intervention staff to allow for examination of the trajectory of weight loss.
Program Satisfaction | 3 months and 6 months
  Program Satisfaction:
  Participants will be asked to complete a program Satisfaction Survey. The Satisfaction Survey is a self-administered survey scored on a 5-point Likert scale.
Program Satisfaction - Open-ended Survey | 6 months
  Program Satisfaction:
  Open-ended Satisfaction Survey. Participants will be asked to complete a Open-ended Satisfaction survey that consist of 2 open-ended questions, and asked respondents to report on their satisfaction with the program.
Change in Weight-related Quality of Life | Baseline, 3 months, and 6 months
  The Impact of Weight on Quality of Life-Lite (IWQOL-Lite) is a validated self-report measure for an individual's perception of how their weight affects their day-to-day life and will be completed at baseline, Months 3 and 6. Respondents rate the degree to which their weight affects them on 31 items using a five-point Likert scale (1, never true; 2, rarely true; 3, sometimes true; 4, usually true; 5, always true). The IWQOL-Lite consists of 5 scales (physical function, self-esteem, sexual life, public distress, and work).
Change in Hunger | Baseline, 3 months, and 6 months
  The most commonly used tool to measure subjective sensations of hunger is the Visual Analogue Scale (VAS). A VAS measures sensations that range across a continuum of values and cannot be easily directly measured. Operationally, the VAS is a horizontal line measuring exactly 100 mm in length, anchored by word descriptors (i.e., Not at all hungry, Extremely hungry) at each end. At baseline, Months 3 and 6, participants will be asked to complete a three item VAS by placing a mark on the line at the point they feel represents their response to the question.

CONTACTS AND LOCATIONS:
Overall Officials: Renee J. Rogers, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No